CLINICAL TRIAL: NCT07195669
Title: Nonopioid Versus Opioid Management of Post-operative Pain Following Oral & Maxillofacial Surgery: A Randomized Controlled Trial
Brief Title: RCT: Suzetrigine vs Norco for Post-op Pain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jacob Lensing (Other)
Responsible Party: Sponsor-Investigator, Jacob Lensing, Resident, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSU8322
Record Dates: First submitted 2025-09-24; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pain Control
Keywords: pain; analgesic; post-operative
MeSH Terms: conditions — Agnosia; Pain | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suzetrigine + Ibuprofen (Experimental): - Group 1 will receive a 100-mg oral loading dose of Journavx (suzetrigine), followed by a 50-mg maintenance dose every 12 hours (the high-dose group) and ibuprofen 800 mg q8h for 72 hours after surgery (1).
  Interventions: Drug: Suzetrigine (SUZ)
- Opioid + Ibuprofen (Active Comparator): - Group 2 will receive ibuprofen 800 mg x 15 tabs q8h scheduled and hydrocodone/acetaminophen 5/325 q8h PRN for 72 hours after surgery. Patients will be informed not to exceed 3g of acetaminophen or 3200 mg ibuprofen (1).
  Interventions: Drug: Norco

INTERVENTIONS:
Drug: Suzetrigine (SUZ) — Used in the course of acute post-operative pain following oral and maxillofacial surgeries
  Arms: Suzetrigine + Ibuprofen
Drug: Norco — Its standard of care
  Arms: Opioid + Ibuprofen

SUMMARY:
Journavx (suzetrigine) is a novel non-opioid analgesic that is FDA approved for acute pain management and may offer a promising alternative for managing postoperative pain. Suzetrigine is selective inhibitor of the sodium channel NaV1.8, for managing acute pain. NaV1.8, a sodium channel, plays a key role in transmitting pain signals. Importantly, this channel is minimally expressed in the brain, enabling effective pain control without the potential central nervous system side effects of respiratory depression and addiction associated with opioids. Clinical trials have shown Journavx to be effective in managing moderate to severe post-operative pain equal to that of opiates. This study aims to further evaluate the efficacy and safety of Journavx in managing post-operative pain after third molar removal and orthognathic surgery.

Participants in this study should be aged 18-45 without significant autoimmune diseases, chronic kidney disease, liver disease, chronic pain disorder including temporomandibular joint disorder, bleeding disorders, pregnant or nursing, undergoing either extraction of both lower third molars or orthognathic surgery of both the maxilla and mandible.

DETAILED DESCRIPTION:
Every year millions of oral and maxillofacial surgical procedures are performed globally, with patients frequently experiencing significant postoperative pain that can persist long after hospital discharge1. One of the most frequent outpatient procedures performed by oral surgeons is third molar extraction, with an estimated 10 million such procedures performed annually in the United States alone2. Orthognathic surgery, another common procedure, has been reported to have the highest postoperative pain scores compared to other oral and maxillofacial procedures3. Inadequate pain control in this critical period can lead to impaired function, slower healing, and may be a factor in prolonged pain in the subacute setting4. Despite the critical importance of effective postoperative pain control to patient recovery, the optimal analgesic approach remains a topic of debate, with both opioid and non-opioid medications utilized in clinical practice5,6.

Opioids have long played a central role in managing postoperative pain in oral surgery7. The risks associated with opioid use are well-documented7,8. Addiction and misuse are the most widely discussed opioid side effects in the public. However, more common side effects, such as nausea, vomiting, constipation, respiratory depression, and sedation, can have a profound effect on morbidity. Furthermore, there is a growing body of evidence suggesting that the overprescription of opioids following common procedures like wisdom tooth extraction contributes to the larger opioid epidemic8. These risks underscore the need for alternative pain management strategies that minimize or eliminate the need for opioids.

Journavx (suzetrigine) is a novel non-opioid analgesic that offers a promising alternative for managing postoperative pain9,10. Suzetrigine is selective inhibitor of the sodium channel NaV1.8, for managing acute pain. NaV1.8, a sodium channel subtype found primarily in peripheral nerves and dorsal root ganglia, plays a key role in transmitting nociceptive signals. Importantly, this channel is minimally expressed in the brain, enabling selective blockade to provide targeted, effective analgesia without the potential central nervous system side effects of respiratory depression and addiction associated with opioids11. Clinical trials have shown Journavx to be effective in managing moderate to severe post-operative pain equal to that of opiates11. This study aims to further evaluate the efficacy and safety of Journavx in managing post-operative pain after third molar removal and orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 years requiring extraction of impacted mandibular bilateral third molar teeth, uncomplicated mesioangular impacted teeth, or vertical impaction of unerupted and impacted mandibular third molars.
* Patients aged 18-45 years undergoing bimaxillary orthognathic surgery.

Exclusion Criteria:

* Pregnant or nursing, history of prior opioid abuse, have history of temporomandibular dysfunction or local myofascial pain disorder preoperatively, with history of congenital syndrome requiring previous surgeries, orthognathic revisions, have a bleeding disorder, cannot receive instruction in English, are currently utilizing analgesics for another painful condition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 72 hours post op
  Numeric Pain Rating Scale (NPRS, a numeric version of a visual-analogue scale; scores range from 0 to 10, with higher scores indicating greater pain) at 8, 16, 24, 36, 48, 72 hours following surgery (6 time points)

SECONDARY OUTCOMES:
Adverse drug effects | 72 hours
  Any unwanted side effects of the medication such as: headaches, nausea, rash, itching, and/or muscle spasms

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lensing, DDS, Principal Investigator — LSUHSC
Locations (1):
- LSU Dental School, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones J, Correll DJ, Lechner SM, Jazic I, Miao X, Shaw D, Simard C, Osteen JD, Hare B, Beaton A, Bertoch T, Buvanendran A, Habib AS, Pizzi LJ, Pollak RA, Weiner SG, Bozic C, Negulescu P, White PF; VX21-548-101 and VX21-548-102 Trial Groups. Selective Inhibition of NaV1.8 with VX-548 for Acute Pain. N Engl J Med. 2023 Aug 3;389(5):393-405. doi: 10.1056/NEJMoa2209870. PMID 37530822
- [Background] Mutlu I, Abubaker AO, Laskin DM. Narcotic prescribing habits and other methods of pain control by oral and maxillofacial surgeons after impacted third molar removal. J Oral Maxillofac Surg. 2013 Sep;71(9):1500-3. doi: 10.1016/j.joms.2013.04.031. PMID 23948362
- [Background] Mobini A, Mehra P, Chigurupati R. Postoperative Pain and Opioid Analgesic Requirements After Orthognathic Surgery. J Oral Maxillofac Surg. 2018 Nov;76(11):2285-2295. doi: 10.1016/j.joms.2018.05.014. Epub 2018 May 19. PMID 29886112
- [Background] Sancho-Puchades M, Valmaseda-Castellon E, Berini-Aytes L, Gay-Escoda C. Quality of life following third molar removal under conscious sedation. Med Oral Patol Oral Cir Bucal. 2012 Nov 1;17(6):e994-9. doi: 10.4317/medoral.17677. PMID 22926461
- [Background] Tuzuner AM, Ucok C, Kucukyavuz Z, Alkis N, Alanoglu Z. Preoperative diclofenac sodium and tramadol for pain relief after bimaxillary osteotomy. J Oral Maxillofac Surg. 2007 Dec;65(12):2453-8. doi: 10.1016/j.joms.2007.06.622. PMID 18022468
- [Background] Park R, Mohiuddin M, Arellano R, Pogatzki-Zahn E, Klar G, Gilron I. Prevalence of postoperative pain after hospital discharge: systematic review and meta-analysis. Pain Rep. 2023 May 8;8(3):e1075. doi: 10.1097/PR9.0000000000001075. eCollection 2023 May-Jun. PMID 37181639